CLINICAL TRIAL: NCT04843631
Title: Bioequivalence Randomised, Double-blind, 3-parallel -Group Phase I Study of BFI-751 Compared With EU-STELARA® and US-STELARA® in Healthy Adult Volunteers
Brief Title: Bioequivalence Phase I Study of BFI-751 Compared With EU and US-STELARA® in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioFactura Australia Pty Ltd. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BFTA-AU-001
Record Dates: First submitted 2021-03-23; First posted 2021-04-13 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, parallel group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double-blinded. Sealed participant-specific code break envelopes will be produced by the unblinded statistician so that the treatment assigned to each participant can be obtained if required, in an emergency only, where knowledge of the randomisation code is required to provide appropriate treatment. The code break envelopes will be retained at the clinical unit in a secure, accessible location. Those blinded to study drug assignment include the sponsor, the PI, clinical study personnel participating in participants' care or clinical evaluations, and the study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: BFI-751 (Experimental): On Day 1, participants will be randomised to receive a single SC dose of 45 mg/0.5mL BFI-751
  Interventions: Drug: BFI-751
- Arm B: EU-STELARA® (Active Comparator): On Day 1, participants will be randomised to receive a single SC dose of 45 mg/0.5mL EU- STELARA®
  Interventions: Drug: EU-STELARA®
- Arm C: US-STELARA®. (Active Comparator): On Day 1, participants will be randomised to receive a single SC dose of 45 mg/0.5mL US- STELARA®
  Interventions: Drug: US-STELARA®

INTERVENTIONS:
Drug: BFI-751 — Single use vial, solution
  Other Names: Ustekinumab Biosimilar
  Arms: Arm A: BFI-751
Drug: EU-STELARA® — Pre-filled syringe, solution
  Other Names: STELARA® (ustekinumab)
  Arms: Arm B: EU-STELARA®
Drug: US-STELARA® — Pre-filled syringe, solution
  Other Names: STELARA® (ustekinumab)
  Arms: Arm C: US-STELARA®.

SUMMARY:
BFI-751 is being developed by BioFactura Australia Pty Ltd as a biosimilar drug to Stelara® (EU licenced and US licenced) (ustekinumab) is a prescription biologic medicine used to treat people with Crohn's disease, Ulcerative Colitis, plaque psoriasis and psoriatic arthritis. Stelara® is an immune suppressant that reduces the effects of inflammatory proteins within the body.

This is the first time BFI-751 will be given to humans. The primary purpose of this study is to compare the pharmacokinetics (the study of what the body does to the drug, referring to the movement of any drug going into, through, and out of the body) by checking to see if the blood levels of 751-BFI are comparable with US-Stelara® and EU-Stelara® following a single injection under the skin.

The secondary purposes of this study are:

* to assess the safety of BFI-751,
* study how well the healthy volunteers tolerate it and
* to also assess the immune response to it in healthy volunteers.

DETAILED DESCRIPTION:
This is a two centre, bioequivalence, randomized, double-blind, 3 parallel group Phase 1 study of BFI-751 compared with EU-Stelara ® and US-Stelara ® in healthy adult volunteers.

Within 28 days of screening, eligible participants will commence a confinement period on Day -1. The participants will receive a 45mg dose of either BFI-751, Stelara-US ® or Stelara-EU® in a blinded manner on Day 1 and will remain in the clinic until Day 2.

Participants will then return to the clinic as outpatients on Days 3, 5, 8, 11, 15, 22, 29, 36, 43,57, 71 and 85 for safety assessments.

A total of up to 228 eligible participants will be enrolled and randomised in a 1:1:1 ratio (BFI-751: EU-Stelara ® : US-Stelara ® ).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will be included in the study if they meet all of the following criteria at screening, and after check-in on Day -1, prior to dose administration:

  1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
  2. Adult male and female volunteers, 18 to 50 years of age (inclusive).
  3. Subjects who smoke no more than 2 cigarettes or equivalent per week can be included in the study but must be willing to abstain from smoking 7 days prior to admission and during the confinement period. Subjects must have a negative test for cotinine prior to check-in on Day -1.
  4. Body mass index (calculated) within the range of 18 to 32 kg/m2 inclusive.
  5. Body weight ≥ 50 kg and ≤ 100 kg inclusive.
  6. Medically healthy without clinically significant abnormalities, including:

     1. Physical examination without any clinically significant findings, in the opinion of the Investigator.
     2. Systolic blood pressure (BP) in the range of 90 to 145 mm Hg (inclusive) and diastolic BP in the range of 50 to 90 mm Hg (inclusive) after at least 5 minutes in the supine position.
     3. Heart rate (HR) in the range of 40 to 100 beats/min (inclusive) after at least 5 minutes rest in a supine position.
     4. Normal body temperature 35.5 to 37.7°C (inclusive).
     5. Triplicate 12-lead electrocardiogram (ECG), taken after the volunteer has been supine for at least 5 minutes, with a QT interval corrected using the Fridericia method (QTcF) ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities, in the opinion of the Investigator.
     6. No clinically significant findings in serum chemistry, haematology, coagulation and urinalysis examinations, in the opinion of the Investigator.

     Assessments may be repeated once, if abnormal values were recorded in the first instance, at the discretion of the Investigator.
  7. Female volunteers must:

     1. Be of non-child-bearing potential i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the Screening visit) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone level indicative of postmenopausal status per local laboratory definition), OR
     2. If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant, and, if engaging in sexual intercourse with a male partner must agree to use an acceptable method of contraception for from signing the consent form until at least 15 weeks after the last dose of study drug.
  8. Male volunteers, must agree not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable form of contraception from signing the consent form until at least 15 weeks after the last dose of study drug.
  9. Have suitable venous access for blood sampling.
  10. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

* Healthy volunteers will be excluded from the study if there is evidence of any of the following at screening or after check-in on Day -1, prior to dose administration:

  1. 1. Prior exposure to STELARA® (Ustekinumab).
  2. Have a history of hypersensitivity or allergic reactions (either spontaneous or following drug administration) to any of the active or formulation ingredients of the study treatments components.
  3. Have a history of or presence of disease determined by the PI to be clinically significant including:

     1. gastrointestinal (including diverticulitis, stomach ulcers, inflammatory intestinal disease, gastrointestinal perforations/fistulae/intra-abdominal abscess).
     2. any other internal, non-gastrointestinal fistulae that is at an increased risk of bleeding.
     3. haematological (including pancytopenia, aplastic anaemia or blood dyscrasia).
     4. renal, hepatic, pulmonary, neurologic, psychiatric, metabolic (including known diabetes mellitus), or
     5. allergic disease excluding mild asymptomatic seasonal allergies.
  4. Have a history of prolonged immunosuppressant therapy, or photochemotherapy treatment.
  5. Presence or evidence of recent sunburn, scar tissue, tattoo (more than 25% of body area), open sore or branding that, in the opinion of the Investigator, would interfere with interpretation of skin adverse reactions.
  6. Have a history of and/or current cardiac disease defined as one of the following:

     1. History of congestive heart failure; angina pectoris requiring anti-anginal medication.
     2. Evidence of transmural infarction on ECG.
     3. History of sustained hypertension (systolic > 180 mmHg and/or diastolic > 100 mmHg) or hypertensive crisis or hypertension encephalopathy.
     4. Clinically significant valvular heart disease, or severe arterial thromboembolic events.
  7. Have a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus, human immunodeficiency virus (HIV) or history of active, latent or inadequately treated tuberculosis (TB) infection.
  8. Positive serum pregnancy test for women of childbearing potential at the Screening visit or positive urine pregnancy test with confirmatory serum pregnancy test prior to dosing on Day 1.
  9. Females who are breastfeeding.
  10. Have a history of cancer including lymphoma, leukaemia and skin cancer (volunteers with a maximum of 1 surgically resected basal cell carcinoma or squamous cell carcinoma are permitted).
  11. Have an illness within 30 days prior to screening, or prior to dosing, that is classed as clinically significant by the Investigator.
  12. Prior exposure to any investigational monoclonal antibody within 12 months or 5 half-lives of the previous drug (if known), whichever is longer, prior to study drug administration.
  13. Have participated in another clinical study of an investigational drug (excluding monoclonal antibody) within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to the administration of the study drug, or are currently participating in another clinical study of an investigational drug, or intending to participate in another clinical study of an investigational drug before completion of all scheduled evaluations in this clinical study.
  14. Any clinically significant infection, in the opinion of the Investigator, ongoing at screening or admission to the clinical unit.
  15. Have had major surgery within 30 days prior to screening or will have an operation between screening and the end of study visit, or have any unhealed wound, including wound dehiscence and wound healing complications requiring medical intervention.
  16. Have received any vaccine(s) within 14 days prior to check in on Day -1, or is planning to receive any vaccine with 14 days following dose administration on Day 1.
  17. Have received a Bacillus Calmette-Guerin (BCG) vaccination within 1 year prior to dose administration, or is planning to receive a BCG vaccination within 1 year following dose administration.
  18. History of alcohol abuse (defined as more than 12 standard drinks per week or more than 4 standard drinks on > 3 days per week; where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], 30 mL spirit [40% Alc./Vol]) within 12 weeks prior to the screening visit.
  19. Positive drug or alcohol test results. In the event the urinary drug test is positive, the test may be repeated once (at the discretion of the PI) to confirm eligibility.
  20. Have donated > 100 mL blood within 4 weeks prior to the administration of the study drug.
  21. Abnormal or irregular bowel movements, in the opinion of the Investigator.
  22. Any history of non-traumatic haemorrhage (i.e. any haemorrhage requiring medical intervention) or any condition which may increase bleeding risk including clotting disorders, thrombocytopenia (platelet count < 150, 000 per μL) or an international normalised ratio higher than 1.5.
  23. Impaired liver function as determined by a serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)> 1.5 x upper limit of normal (ULN) at screening or admission. Subjects with values between ULN and 1.5 x ULN may be included in the study if considered not clinically significant by the Investigator.
  24. Use of any prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, which, in the opinion of the Investigator, could affect the outcome of the study. The following exceptions apply:

      1. Contraceptives for WOCBP are permitted.
      2. Paracetamol (up to a maximum of 4 doses of 500 mg per day, and no more than 3g per week) is permitted.
      3. Ibuprofen (up to a maximum of 4 doses of 200 mg per day) is permitted.
  25. Consumption of any foods containing poppy seeds within 48 hours prior to screening and admission to the clinical centre.
  26. Presence of proteinuria (other than trace amounts i.e., +, ++/+++).
  27. Personal history of venous thromboembolic events or idiopathic venous thromboembolic events in a first degree relative.
  28. Any person who is an employee of an Investigator or Sponsor, or an immediate relative of an Investigator.
  29. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence- Cmax | From Baseline to Day 85
  Compare Maximum observed concentration (Cmax) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection
Bioequivalence-Tmax | From Baseline to Day 85
  Compare Time to Cmax (Tmax) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection
Bioequivalence - Area under the concentration-time curve from time zero to the last measurable concentration (AUC0-tlast) | From Baseline to Day 85
  Compare Area under the concentration-time curve from time zero to the last measurable concentration (AUC0-tlast) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection
Bioequivalence - Total AUC after extrapolation from time t to time infinity (AUC0-inf) | From Baseline to Day 85
  Compare Total AUC after extrapolation from time t to time infinity (AUC0-inf) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection
BioEquivalence - Elimination rate constant (Kel) | From Baseline to Day 85
  Compare Elimination rate constant (Kel) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection
Bioequivalence - Apparent terminal elimination half-life (t1/2) | From Baseline to Day 85
  Compare Apparent terminal elimination half-life (t1/2) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection
Bioequivalence - Volume of distribution (Vz) | From Baseline to Day 85
  Compare Volume of distribution (Vz) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection
Bioequivalence - Apparent clearance (CL) | From Baseline to Day 85
  Compare Apparent clearance (CL) of BFI-751 with EU-Stelara and US-Stelara following a single 45 mg SC injection

SECONDARY OUTCOMES:
Safety and tolerability - Incidence, type and severity of Adverse Events | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Incidence, type and severity of Adverse Events
Safety and tolerability - Changes from baseline in clinical laboratory results (haematology, serum chemistry, coagulation, and urinalysis) | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Changes from baseline in clinical laboratory results (haematology, serum chemistry, coagulation, and urinalysis)
Changes from baseline in vital signs parameter - systolic and diastolic blood pressure in mmHg | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Changes from baseline in vital signs parameter - systolic and diastolic blood pressure in mmHg
Changes from baseline in vital signs parameter - heart rate in beats per minute | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Changes from baseline in vital signs parameter - heart rate in beats per minute
Changes from baseline in vital signs parameter - respiratory rate in breaths per minute | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Changes from baseline in vital signs parameter - respiratory rate in breaths per minute
Changes from baseline in vital signs parameter - body temperature in degrees Celsius | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Changes from baseline in vital signs parameter - respiratory rate in breaths per minute
Changes from baseline in physical examination findings - height in centimeters | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Changes from baseline in physical examination findings - height in centimeters. Weight and height will be combined to report BMI in kg/m^2.
Changes from baseline in physical examination findings - weight in kilograms | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Changes from baseline in physical examination findings - weight in centimeters. Weight and height will be combined to report BMI in kg/m^2.
Changes from baseline in triplicate 12-lead electrocardiograms (ECG) Ventricular HR | From Baseline to Day 85
  Measured by assessment of Ventricular HR as normal, not having a clinically significant abnormality or having a clinically significant abnormality
Changes from baseline in triplicate 12-lead electrocardiograms (ECG) PR Interval | From Baseline to Day 85
  Measured by assessment of PR interval as normal, not having a clinically significant abnormality or having a clinically significant abnormality
Changes from baseline in triplicate 12-lead electrocardiograms (ECG) RR interval | From Baseline to Day 85
  Measured by assessment of RR interval as normal, not having a clinically significant abnormality or having a clinically significant abnormality
Changes from baseline in triplicate 12-lead electrocardiograms (ECG) QRS duration | From Baseline to Day 85
  Measured by assessment of QRS duration as normal, not having a clinically significant abnormality or having a clinically significant abnormality
Changes from baseline in triplicate 12-lead electrocardiograms (ECG) QT interval | From Baseline to Day 85
  Measured by assessment of QT interval as normal, not having a clinically significant abnormality or having a clinically significant abnormality
Changes from baseline in triplicate 12-lead electrocardiograms (ECG) QTcF | From Baseline to Day 85
  Measured by assessment of QTcF as normal, not having a clinically significant abnormality or having a clinically significant abnormality
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: general appearance
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: head
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: ears
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: eyes
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: nose and throat
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: neck (including thyroid and lymph nodes)
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: respiratory
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: cardiovascular
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: gastrointestinal
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: renal
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: neurological condition
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: musculoskeletal system
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: skin
Occurence of any clinical significant (CS) physical examination findings | From Baseline to Day 85
  Measured by assessment of the following system: any other focused assessments suggested by the presence of specific symptoms.
Safety and Tolerability - Incidence, type and severity of injection site reactions. | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Incidence, type and severity of injection site reactions.
Immunogenicity - incidence of antidrug antibody (ADA) | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Incidence of antidrug antibody (ADA) and/or neutralising antibody (nAb) against 751-BFI, US- and EU-STELARA®, including titres for ADA.
Immunogenicity - incidence of neutralising antibody (nAb) | From Baseline to Day 85
  The secondary objective of the study is to investigate the safety, tolerability and immunogenicity of BFI-751, EU-Stelara and US-Stelara including Incidence of neutralising antibody (nAb) against 751-BFI, US- and EU-STELARA®.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey N Hausfeld, MD, Study Director — BioFactura Australia Pty Ltd.; Kristi McLendon, Principal Investigator — Nucleus Network; Emir Redzepagic, Principal Investigator — CMAX; Christian Schwabe, Principal Investigator — NZCR
Locations (3):
- Australia (2):
  - Nucleus Network, Brisbane, Queensland
  - CMAX, Adelaide, South Australia
- NZCR, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hausfeld JN, Challand R, McLendon K, Macapagal N, Bruce-Staskal P, Fiaschetti C, Sampey DB. Pharmacokinetic Profiles of a Proposed Biosimilar Ustekinumab (BFI-751): Results From a Randomized Phase 1 Trial. Clin Pharmacol Drug Dev. 2023 Oct;12(10):1001-1012. doi: 10.1002/cpdd.1305. Epub 2023 Jul 22. PMID 37483071